CLINICAL TRIAL: NCT00130858
Title: a Multicenter Clinical Trial for the Treatment of Children and Adolescents With Soft Tissue Sarcoma Stage 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cooperative Weichteilsarkom Study Group (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWS-IV 2002
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Topotecan; Carboplatin

INTERVENTIONS:
Drug: Topotecan
Drug: Carboplatin

SUMMARY:
Phase II Study to evaluate the response on two blocks of topotecan and carboplatin

DETAILED DESCRIPTION:
Phase II study for patients with chemosensible soft tissue sarcoma stage IV in children and adolescents ; response according to RECIST criteria following two blocks of combination therapy consisting of Topotecan and carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Soft tissue sarcoma chemosensible, stage IV
* age < 21
* measurable tumor lesions

Exclusion Criteria:

* Lack of cooperation by the patient
* no willingness of follow-up examinations
* participation on another clinical trial at the same time
* death due to the sickness within four weeks

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Response according to RECIST criteria

SECONDARY OUTCOMES:
Toxicity
Overall-Survival
Event-free-survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klingebiel, Prof. Dr., Study Chair — Klinikum der Johann Wolfgang Goethe-Universität
Locations (38):
- Germany (38):
  - HELIOS Klinikum Erfurt GmbH, Erfurt, Saxony
  - Zentralklinikum, Augsburg
  - Klinikum Berlin-Buch, Berlin
  - Virchow Klinik, Berlin
  - Zentrum für Kinderheilkunde, Bonn
  - Zentralkrankenhaus Bremen, Bremen
  - Klinikum der Stadt Köln, Cologne
  - Universitäts-Kinderklinik, Cologne
  - Universitätsklinik der technischen Universität Dresden, Dresden
  - Heinrich-Heine-Universität, Düsseldorf
  - Universitätsklinik für Kinderund Jugendliche, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum der Universität, Frankfurt
  - Universitäts-Kinderklinik Freiburg, Freiburg im Breisgau
  - Klinikum der Justus-Liebig-Universität, Giessen
  - Georg-August-Universität, Göttingen
  - Universitäts-Kinderklinik Hamburg, Hamburg
  - Kinderklinik der Medizinischen Hochschule, Hanover
  - Universitäts-Kinderklinik, Heidelberg
  - Universitäts-Kinderklinik, Homburg/saar
  - Klinik für Kinder- und Jugendmedizin, Jena
  - Städtisches Klinikum Karlruhe, Karlsruhe
  - Klinikum der Universität Kiel, Kiel
  - Universitätsklinik und Poliklinik, Leipzig
  - Kinderklinik St. Annastift, Ludwigshafen
  - Medizinische Universität zu Lübeck, Lübeck
  - Medizinische Fakultät, Magdeburg
  - Klinikum der Johannes-Gutenberg-Universität, Mainz
  - Dr. von Haunersches Kinderspital, München
  - Städtisches Krankenhaus Technische Universität Schwabing, München
  - Westfälische Wilhelms-Universität, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinik St. Hedwig, Regensburg
  - Johanniter-Kinderklinik, Sankt Augustin
  - Olgahospital, Stuttgart
  - Universitäts-Kinderklinik, Tübingen
  - Universitäts-Kinderklinik, Ulm
  - Universitäts-Kinderklinik, Würzburg